CLINICAL TRIAL: NCT01419054
Title: Understanding Hand Hygiene Behavior at Unidad Nacional Oncologia Pediatrica: A Focus Group Approach
Brief Title: Understanding Hand Hygiene Behavior at Unidad Nacional Oncologia Pediatrica
Acronym: HHFG
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HHFG
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Hand Hygiene Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Healthcare associated infections increase morbidity and mortality among all hospitalized patients, especially in those who are immunocompromised, in both developed and in countries with limited resources. However, when resources are limited, infection prevention and control measures are often overlooked by personnel and institutions. Hand hygiene has been shown numerous times to be the most effective way to prevent infections in the healthcare setting. In Unidad Nacional de Oncologia Pediatrica (UNOP) in Guatemala City, Guatemala, there have been several infrastructural improvements and periodic education and promotion activities. Still, acceptable hand hygiene compliance has not yet been sustainably achieved. The investigators wish to study reasons why staff at UNOP do or do not practice hand hygiene when it is indicated through the use of focus groups and interviews.

DETAILED DESCRIPTION:
Healthcare associated infections (HAI) are a concern in all parts of the world. Patients who are immune-compromised by chemotherapy, HIV/AIDS, or organ transplant are especially susceptible to infection. In addition to the opportunistic infections that these patients are at risk of acquiring, the emergence of methicillin resistant Staphylococcus aureus and vancomycin resistant Enterococcus species pose a risk to healthy individuals as well. Hand hygiene is one of the most important infection prevention practices for everyone in a hospital. In resource-poor countries, infection prevention and control programs are often neglected due to a lack of funding and organizational priorities. The Division of Infectious Diseases - International Outreach (ID-IO) has partnered with several hospitals in Latin America to mentor healthcare providers and provide key supplies so that they deliver the best care and prevent infection in units where the patients have the greatest risk of acquiring and dying from infections. Because of its importance, ID-IO has focused on hand hygiene as a building block for safe care at these hospitals; therefore, each year, at these hospitals, a hospital-wide education and promotion effort on hand hygiene is completed. The topics covered are general hospital hygiene, access to hand hygiene stations, and ensuring that adequate supplies for hand hygiene are available. Observation of hand hygiene practices before, during, and after bedside clinical activities shows there is a temporary improvement in compliance with current hand hygiene guidelines; however, the rates of compliance decline again as HAIs increase. In this study, the investigators propose to use already available hand hygiene practice surveillance and healthcare associated infection documentation and obtain the healthcare professionals' opinions and experiences that affect the practice of hand hygiene. Because motivation and barriers to practice hand hygiene derive from more than just education and adequate supplies, the investigators would like to understand the reasons why the healthcare providers do and do not practice hand hygiene when indicated. The methods to be used in this study are focus group meetings and structured interviews with staff of Unidad Nacional de Oncologia Pediatrica in Guatemala City, Guatemala.

ELIGIBILITY:
Inclusion Criteria:

* Position held/job responsibilities of staff at Unidad Nacional de Oncologia Pediatrica in Guatemala City, Guatemala.

Exclusion Criteria:

* Does not hold position or have job responsibilities at Unidad Nacional de Oncologia Pediatrica in Guatemala City, Guatemala.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health-care providers
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Identify changes, if any, in hand hygiene following improvements identified during the focus group sessions aimed at increasing hand hygiene compliance of staff members. | One (1) year
  The investigators propose to use already available hand hygiene practice surveillance and healthcare-associated infection documentation and obtain the healthcare professionals' opinions and experiences that affect the practice of hand hygiene to assess: (1) hand hygiene education and promotion; (2) access to hand hygiene supplies at the point of care; and (3) in other specific barriers to practice hand hygiene.

SECONDARY OUTCOMES:
Identify educational, motivational, and infrastructural issues that need to be addressed to increase hand hygiene practice compliance. | One (1) year
  Focus group meetings and structured interviews with staff with be used to assess the issues to be addressed.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M. Johnson, PhD, Study Chair — St. Jude Children's Research Hospital
Locations (1):
- Unidad Nacional Oncologia Pediatrica, Guatemala City, Departamento de Guatemala, Guatemala

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org